CLINICAL TRIAL: NCT01349127
Title: Randomised Placebo-controlled Supplementation Study With Vitamin D and Calcium in Breastfeeding Mothers
Brief Title: Trial to Assess Vitamin D Requirements in Lactating Women
Acronym: DMUMs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: Irish Government Department of Agriculture, Food and Fisheries, Ireland (Unknown)
Responsible Party: Principal Investigator, Mairead Kiely PhD, Professor of HUman Nutrition, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Cork Vitamin D 06/RD/C/533
Record Dates: First submitted 2011-04-21; First posted 2011-05-06 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Vitamin D Deficiency; Vitamin D Insufficiency
Keywords: Vitamin D; Cholecalciferol; Nutrient requirements; Randomised Controlled Trial; Lactation; pregnancy; Cord blood; Human milk; serum 25-hydroxyvitamin D; deficiency; insufficiency; nutrition
MeSH Terms: conditions — Vitamin D Deficiency; Breast Feeding | interventions — Cholecalciferol; Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 20µg Vitamin D3 (Active Comparator): Arm will receive per day one gelatin capsule containing 20µg (800IU) of vitamin D3 (Cholecalciferol).
  Interventions: Dietary Supplement: 20µg Vitamin D3
- 20µg Vitamin D3 + 500 mg Calcium (Active Comparator): Arm will receive per day one gelatin capsule containing 20µg (800IU) of vitamin D3 (Cholecalciferol) and one tablet of calcium carbonate containing 500mg of calcium.
  Interventions: Dietary Supplement: 20µg Vitamin D3 + 500 mg Calcium
- Placebo (Placebo Comparator): Arm will receive one gelatin capsule containing 0µg (0IU) of vitamin D3 (Cholecalciferol).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 20µg Vitamin D3 — 20µg (800IU) of vitamin D3/day for 12-weeks while lactating, commencing 10-14 days post-partum.
  Other Names: Cholecalciferol
  Arms: 20µg Vitamin D3
Dietary Supplement: 20µg Vitamin D3 + 500 mg Calcium — 20µg (800IU) of vitamin D3 + 500mg calcium carbonate/day for 12-weeks while lactating, commencing 10-14 days post-partum.
  Other Names: Cholecalciferol and Calcium
  Arms: 20µg Vitamin D3 + 500 mg Calcium
Dietary Supplement: Placebo — One gelatin placebo capsule containing zero vitamin D3 taken for 12-weeks while lactating, commencing 10-14 days post-partum.
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled trial of vitamin D supplementation with 20mcg cholecalciferol (to achieve a total intake of 25mcg/day), with or without 500mg calcium to assess vitamin D requirements in lactating women and to ascertain whether vitamin D supplementation at levels sufficient to achieve defined thresholds of maternal serum 25-hydroxyvitamin D will increase the vitamin D content of maternal milk. The study will also report serum 25-hydroxyvitamin D in maternal-cord dyads over a 12-month period and describe the relationship between them. Information on maternal iPTH levels, anthropometry, diet and sun exposure will also be reported.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women intending to breast feed their infant for at least 12-weeks
* Pregnant women >20 weeks gestation
* Pregnant women >18 years of age
* Pregnant women in good general health

Exclusion Criteria:

* Consumption of a vitamin D-containing supplement(>10µg/day) in the 3 months prior to commencing the trial
* Consumption of a vitamin D or calcium containing supplement during the 12- week trial
* Mothers taking a vacation to a sunny climate or using a solarium during the 12-week trial
* Mothers with pre-existing type 1 or type 2 diabetes
* Mothers with pre-existing hypertension
* Mothers with diagnosed hypercalcemia
* Mothers with diagnosed intestinal malabsorption conditions
* Mothers with multiple fetuses (e.g. twins)
* Consumption of medications known to interfere with vitamin D metabolism.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Serum 25-hydroxyvitamin D in mothers and levels of vitamin D in maternal milk | 12 weeks
  Baseline and endpoint serum 25(OH)D analysis in mothers (week 0 and week 12); baseline, week 4, week 8 and enpoint analysis of vitamin D3, D2 and 25(OH)D in expressed breast milk (hindmilk samples)

SECONDARY OUTCOMES:
Maternal serum iPTH | 12 weeks
  Baseline and endpoint PTH will be measured in mothers

CONTACTS AND LOCATIONS:
Overall Officials: Mairead E Kiely, PhD, Principal Investigator — University College Cork
Locations (1):
- School of Food & Nutritional Sciences, University College Cork,, Cork, Ireland

REFERENCES:
- [Background] Seamans KM, Hill TR, Wallace JM, Horigan G, Lucey AJ, Barnes MS, Taylor N, Bonham MP, Muldowney S, Duffy EM, Strain JJ, Kiely M, Cashman KD. Cholecalciferol supplementation throughout winter does not affect markers of bone turnover in healthy young and elderly adults. J Nutr. 2010 Mar;140(3):454-60. doi: 10.3945/jn.109.113480. Epub 2010 Jan 20. PMID 20089776
- [Background] Hill TR, Cotter AA, Mitchell S, Boreham CA, Dubitzky W, Murray L, Strain JJ, Flynn A, Robson PJ, Wallace JM, Kiely M, Cashman KD. Vitamin D status and parathyroid hormone relationship in adolescents and its association with bone health parameters: analysis of the Northern Ireland Young Heart's Project. Osteoporos Int. 2010 Apr;21(4):695-700. doi: 10.1007/s00198-009-0959-1. Epub 2009 May 13. PMID 19436930
- [Background] Cashman KD, Wallace JM, Horigan G, Hill TR, Barnes MS, Lucey AJ, Bonham MP, Taylor N, Duffy EM, Seamans K, Muldowney S, Fitzgerald AP, Flynn A, Strain JJ, Kiely M. Estimation of the dietary requirement for vitamin D in free-living adults >=64 y of age. Am J Clin Nutr. 2009 May;89(5):1366-74. doi: 10.3945/ajcn.2008.27334. Epub 2009 Mar 18. PMID 19297462
- [Background] Cashman KD, Hill TR, Lucey AJ, Taylor N, Seamans KM, Muldowney S, Fitzgerald AP, Flynn A, Barnes MS, Horigan G, Bonham MP, Duffy EM, Strain JJ, Wallace JM, Kiely M. Estimation of the dietary requirement for vitamin D in healthy adults. Am J Clin Nutr. 2008 Dec;88(6):1535-42. doi: 10.3945/ajcn.2008.26594. PMID 19064513
- [Background] O'Riordan MN, Kiely M, Higgins JR, Cashman KD. Prevalence of suboptimal vitamin D status during pregnancy. Ir Med J. 2008 Sep;101(8):240, 242-3. PMID 18990953
- [Background] Hill TR, McCarthy D, Jakobsen J, Lamberg-Allardt C, Kiely M, Cashman KD. Seasonal changes in vitamin D status and bone turnover in healthy Irish postmenopausal women. Int J Vitam Nutr Res. 2007 Sep;77(5):320-5. doi: 10.1024/0300-9831.77.5.320. PMID 18453316
- [Background] Cashman KD, Hill TR, Cotter AA, Boreham CA, Dubitzky W, Murray L, Strain J, Flynn A, Robson PJ, Wallace JM, Kiely M. Low vitamin D status adversely affects bone health parameters in adolescents. Am J Clin Nutr. 2008 Apr;87(4):1039-44. doi: 10.1093/ajcn/87.4.1039. PMID 18400729
- [Background] Hill TR, Cotter AA, Mitchell S, Boreham CA, Dubitzky W, Murray L, Strain JJ, Flynn A, Robson PJ, Wallace JM, Kiely M, Cashman KD. Vitamin D status and its determinants in adolescents from the Northern Ireland Young Hearts 2000 cohort. Br J Nutr. 2008 May;99(5):1061-7. doi: 10.1017/S0007114507842826. Epub 2008 Jan 15. PMID 18197989
- [Background] Andersen R, Molgaard C, Skovgaard LT, Brot C, Cashman KD, Jakobsen J, Lamberg-Allardt C, Ovesen L. Pakistani immigrant children and adults in Denmark have severely low vitamin D status. Eur J Clin Nutr. 2008 May;62(5):625-34. doi: 10.1038/sj.ejcn.1602753. Epub 2007 Apr 18. PMID 17440527
- [Background] McCarthy D, Collins A, O'Brien M, Lamberg-Allardt C, Jakobsen J, Charzewska J, Kiely M, Flynn A, Cashman KD. Vitamin D intake and status in Irish elderly women and adolescent girls. Ir J Med Sci. 2006 Apr-Jun;175(2):14-20. doi: 10.1007/BF03167942. PMID 16872022
- [Background] Hill TR, O'Brien MM, Lamberg-Allardt C, Jakobsen J, Kiely M, Flynn A, Cashman KD. Vitamin D status of 51-75-year-old Irish women: its determinants and impact on biochemical indices of bone turnover. Public Health Nutr. 2006 Apr;9(2):225-33. doi: 10.1079/phn2005837. PMID 16571177
- [Background] Hill TR, Flynn A, Kiely M, Cashman KD. Prevalence of suboptimal vitamin D status in young, adult and elderly Irish subjects. Ir Med J. 2006 Feb;99(2):48-9. PMID 16548220
- [Background] Andersen R, Molgaard C, Skovgaard LT, Brot C, Cashman KD, Chabros E, Charzewska J, Flynn A, Jakobsen J, Karkkainen M, Kiely M, Lamberg-Allardt C, Moreiras O, Natri AM, O'brien M, Rogalska-Niedzwiedz M, Ovesen L. Teenage girls and elderly women living in northern Europe have low winter vitamin D status. Eur J Clin Nutr. 2005 Apr;59(4):533-41. doi: 10.1038/sj.ejcn.1602108. PMID 15714215
- [Background] Hill T, Collins A, O'Brien M, Kiely M, Flynn A, Cashman KD. Vitamin D intake and status in Irish postmenopausal women. Eur J Clin Nutr. 2005 Mar;59(3):404-10. doi: 10.1038/sj.ejcn.1602088. PMID 15674302
- [Background] Hill TR, O'brien MM, Cashman KD, Flynn A, Kiely M. Vitamin D intakes in 18-64-y-old Irish adults. Eur J Clin Nutr. 2004 Nov;58(11):1509-17. doi: 10.1038/sj.ejcn.1602001. PMID 15138462
- [Background] Muldowney S, Lucey AJ, Paschos G, Martinez JA, Bandarra N, Thorsdottir I, Cashman KD, Kiely M. Relationships between vitamin D status and cardio-metabolic risk factors in young European adults. Ann Nutr Metab. 2011;58(2):85-93. doi: 10.1159/000324600. Epub 2011 Apr 8. PMID 21474925
- [Background] Barnes MS, Horigan G, Cashman KD, Hill TR, Forsythe LK, Lucey AJ, McSorley EM, Kiely M, Bonham MP, Magee PJ, Strain JJ, Wallace JM. Maintenance of wintertime vitamin D status with cholecalciferol supplementation is not associated with alterations in serum cytokine concentrations among apparently healthy younger or older adults. J Nutr. 2011 Mar;141(3):476-81. doi: 10.3945/jn.110.131516. Epub 2011 Jan 26. PMID 21270359
- [Background] Muldowney S, Kiely M. Vitamin D and cardiometabolic health: a review of the evidence. Nutr Res Rev. 2011 Jun;24(1):1-20. doi: 10.1017/S0954422410000259. Epub 2010 Dec 1. PMID 21118613
- See also: Vitamin D Research group at University College Cork — http://www.ucc.ie/en/vitamind/